CLINICAL TRIAL: NCT05179850
Title: Computer Aided Diagnostic Tool on Computed Tomography Images for Diagnosis of Retroperitoneal Tumor in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuhan Yang, Associate Professor, West China Hospital
Other Study IDs: HX-2021477
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Wilms' Tumor; Neuroblastoma; Teratoma; Lymphoma; Sarcoma; Germ Cell Tumor
MeSH Terms: conditions — Wilms Tumor; Neuroblastoma; Teratoma; Lymphoma; Sarcoma; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The internal cohort was retrospectively enrolled in West China Hospital, Sichuan University from June 2010 and December 2020. It is a training and internal validation cohort.
  Interventions: Diagnostic Test: Radiomic Algorithm
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is a external validation cohort.
  Interventions: Diagnostic Test: Radiomic Algorithm

INTERVENTIONS:
Diagnostic Test: Radiomic Algorithm — Different radiomic, machine learning, and deep learning strategies for radiomic features extraction, sorting features and model constriction.

SUMMARY:
The aim of this study was to evaluate the diagnostic efficacy of computer aided diagnostic tool for retroperitoneal tumor using machine learning and deep learning techniques on computed tomography images in children.

DETAILED DESCRIPTION:
The retroperitoneal space extends from the lumbar region to the pelvic region and houses vital structures such as the kidney, the ureter, the adrenal glands, the pancreas, the aorta and its branches, the inferior vena cava and its tributaries, lymph nodes, and loose connective tissue meshwork along with fat. This space thus allows the silent growth of primary and metastatic tumors, such that clinical features appear often too late. The therapeutic regimen differs on various types of retroperitoneal tumor in children. It is damaging for pediatric patients to acquire histological specimens through invasive procedures. Hence, an urgent evaluation is absolutely necessary for preoperative diagnosis in such cases via noninvasive approaches. This study is a retrospective-prospective design by West China Hospital, Sichuan University, including clinical data and radiological images. A retrospective database was enrolled for patients with definite histological diagnosis and available computed tomography images from June 2010 and December 2020. The investigators have constructed deep learning and machine learning radiomics diagnostic models on this retrospective cohort and validated it internally. A prospective cohort would recruit infantile patients diagnosed as retroperitoneal tumor since January 2021. The proposed deep learning model would also be validated in this prospective cohort externally. The aim of this study was to evaluate the diagnostic efficacy of computer aided diagnostic tool for retroperitoneal tumor using machine learning and deep learning techniques on computed tomography images in children.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 18 years old
* Receiving no treatment before diagnosis
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Unavailable computed tomography images
* Without written informed consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who had retroperitoneal tumor and completed the abdominal computed tomography examination before operation, biopsy, neoadjuvant chemotherapy, and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological tumor diagnosis | Baseline
  The diagnosis is defined by histopathological specimens from surgery and/or biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No